CLINICAL TRIAL: NCT04077593
Title: Evaluation de la précision d'Une Mesure téléphonique de la fréquence Respiratoire à l'Aide d'Une Application Mobile - The OPERA Study (On the PhonE Respiratory rAte)
Brief Title: On the PhonE Respiratory rAte Study (OPERA)
Acronym: OPERA
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC18.181; n°IDRCB: 2018-A02039-46 (Other: ID RCB)
Record Dates: First submitted 2018-10-22; First posted 2019-09-04 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Respiratory Rate
Keywords: Respiratory Rate; Telemedicine; Dyspnea; Emergencies
MeSH Terms: conditions — Dyspnea; Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: RRate Mobile app — Test respiratory rate with RRate application

SUMMARY:
Introduction. The increasing use of telephone medical advice requires the development of telemedicine tools to assess the patient's severity. Respiratory rate (RR) is a simple vital parameter and is often associated with morbidity and mortality of patients. There is no standardized measure of RR by telephone.

Objective: The investigators wanted to evaluate the RR measurement by phone using a smartphone application called RRate.

Methods. Adults who have been admitted for less than 6 hours to the emergency department after calling Center 15 and whose main reason for consultation is dyspnea will be included. Patients with non-invasive or tracheotomized ventilation will be excluded. The main objective will be to compare by Bland-Altman method the accuracy of the RRate measurement by phone to a one-minute RR measurement at patient's bedside. Secondary endpoints will evaluate the length of RR measurement according to the different methods used; measurement failure criteria; the accuracy of different measurement techniques (RRate at patient's bedside, impedancemetry, traditional measurement during 15s or 30s).

Expected Results. The accuracy of the RR measurement by RRate over the telephone should be within the limits of agreement. The measurement time should be shorter with the RRate application than with traditional methods. However, the measurement by telephone should not always be feasible in patients with mild dyspnea or with poorly audible breathing.

ELIGIBILITY:
Inclusion Criteria:

* Age >18yo
* Dyspnea as main reason for consultation
* Regulated by "Centre 15"
* Admitted for less than 6hours at emergency department

Exclusion Criteria:

* Non invasive or tracheotomized ventilation
* Cognitive impairment
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every adult patient admitted to Grenoble University Hospital's emergency department whose main reason for consultation is dyspnea and who's been dispatched by "Centre 15"
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-10-21 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
RRate app on the phone precision | 1 minute
  To compare withBland-Altman analysis the accuracy of the RRate measurement by phone to a one-minute respiratory rate measurement at patient's bedside

SECONDARY OUTCOMES:
Efficiency | 1 minute
  length of RR measurement according to the different methods used
Measurement failure criteria by different Rrate methods (by phone, next to the patient and the reference method) | 1 minute
  Wether coughing, talking during measurement, phone hold by another person, has an impact on measurement possibility. The gap between the measurement by different RRate methods (by phone, next to the patient and the reference method)
Accuracy | 1 minute
  Bland Altman analysis : between one minute measurement at patient's bedside and other measurements : RRate app at patient's bedside, impedancemetry, traditional measurement during 15 seconds or 30 seconds
Clinical impact | 1 minute
  qSOFA (sequential Organ Failure Assesment score) obtained with different measurement of the RRate at 60 second
Reproducibility | 1 minute
  Coefficient of variation and Intra-class correlation, of respiratory rate measured twice with : RRate app on the phone, RRate app at patient's bedside, 15 seconds measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Maxime MD Maignan, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Grenoble University Hospital, La Tronche, Isere, France

IPD SHARING:
Plan to Share IPD: No